CLINICAL TRIAL: NCT02971982
Title: Velcade/Dexamethasone/Cyclophosphamide(PCD) Versus Rituximab /Dexamethasone/Cyclophosphamide(RCD) for the Treatment of Patients With Waldenstrom's Macroglobulinemia
Brief Title: PCD Versus RCD for the Treatment of Patients With Waldenstrom's Macroglobulinemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: myeloma-02
Record Dates: First submitted 2016-10-19; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Treatment
MeSH Terms: interventions — Rituximab; Dexamethasone; Cyclophosphamide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rituximab /Dex/CTX (Experimental): rituximab /Dexamethasone/cyclophosphamide 6 cycles followed by rituximab (at least 2 cycles) rituximab:375mg/m2 d1 Dexamethasone:40mg d1-4 cyclophosphamide:750mg/m2,d1-28
  Interventions: Drug: rituximab /Dexamethasone/cyclophosphamide
- Velcade/Dex/CTX (Experimental): Velcade/Dexamethasone/cyclophosphamide 6 cycles followed by velcade (at least 2 cycles) Velcade:1.3mg/m2 d1,d4,d8,d11 Dexamethasone:20mg d1-2,d4-5,d8-9,d11-12 cyclophosphamide:750mg/m2,d1-28
  Interventions: Drug: Velcade/Dexamethasone/cyclophosphamide

INTERVENTIONS:
Drug: rituximab /Dexamethasone/cyclophosphamide — rituximab:375mg/m2 ,Dexamethasone 20mg q12h,cyclophosphamide 750mg
  Arms: rituximab /Dex/CTX
Drug: Velcade/Dexamethasone/cyclophosphamide — Velcade:1.3mg/m2,Dexamethasone 10mg q12h,cyclophosphamide 750mg
  Arms: Velcade/Dex/CTX

SUMMARY:
Patients will receive RCD or PCD combination as induction treatment followed by rituximab or velcade maintenance therapy, as the investigators try to compare the, very good partial remission (VGPR) rate, complete remission (CR) rates, Overall remission rate (MR+CR + VGPR + partial remission (PR) rate), major reaction rate (MRR, PR+VGPR+CR) at the end of the research.

DETAILED DESCRIPTION:
This is an open-label, single-centre, randomised study, looking at a series of 40 patients up to the age of 75 with newly diagnosed Waldenstrom's macroglobulinemia (WM) not previously treated. Patients will receive RCD or PCD combination as induction treatment followed by rituximab or velcade maintenance therapy, as the investigators try to compare the, very good partial remission (VGPR) rate, complete remission (CR) rates, Overall remission rate (MR+CR + VGPR + partial remission (PR) rate), major reaction rate (MRR, PR+VGPR+CR) at the end of the research.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed WM according to the second 2002 WM international working group
* Not previously treated, apart from not regularly received by Chlorambucil
* Aged from 18 to 75 years, both male and female
* Ability to give signed informed consent
* Negative pregnancy test at inclusion (if necessary)
* ECOG from 0 to 2

Exclusion Criteria:

* Known hypersensitivity to rituximab or velcade or cyclophosphamide
* Uncontrolled infection including bacteria, virus and fungus, including active HBV infection
* Organic dysfunction: Bilirubin > 1.5 x normal above, Renal failure requiring dialysis, glutamic pyruvic transaminase (ALT) and Glutamic-Oxaloacetic Aminotransferase (AST) > 2.5 x normal above
* Positive HIV serology
* Serious psychiatric item in the history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Investigators try to compare the very good partial remission (VGPR) rate at the end of the research. | 2 years
Investigators try to compare the complete remission (CR) rates at the end of the research. | 2 years
Investigators try to compare Overall remission rate (MR+CR + VGPR + partial remission (PR) rate) at the end of the research. | 2 years
Investigators try to compare major reaction rate (MRR, PR+VGPR+CR) at the end of the research. | 2 yeas

CONTACTS AND LOCATIONS:
Overall Officials: Fu cheng cheng, Phd, Principal Investigator — First Affiliated Hospital,Soochow University
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No